CLINICAL TRIAL: NCT06674720
Title: Correlation of Site and Size of Adenoid Hypertrophy and Middle Ear Effusion.
Brief Title: It is Accepted That Adenoid Hypertrophy is Related to Otitis Media With Effusion Incidence. Better Understanding of the Correlation Between the Relative Size of AH and the Incidence of Persistent OME May Provide Evidence to Support a More Standardized Approach to the Diagnosis and Treatment of OME.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Abo Alqasem Mohamed Abd Alnaser, Resident, Assiut University
Other Study IDs: Adenoid hypertrophy and MEE
Record Dates: First submitted 2024-09-30; First posted 2024-11-05 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Adenoid Hypertrophy; Middle Ear Effusion
MeSH Terms: conditions — Otitis Media with Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to further investigate the correlation between Site and size of adenoid hypertrophy and middle ear effusion in order to provide evidence for designing a more standardized approach to the diagnosis and treatment of OME.

DETAILED DESCRIPTION:
The adenoid, or the pharyngeal tonsil, is an antibody producing lymphatic tissue located in the superior part of the nasopharynx posteriorly, near the choana and opening of the eustachian tube. They are present from the seventh month of gestation and typically grow until age 5. Adenoid tissue can be found extending to the eustachian tube opening and the fossa of Rosenmuller. The fossa of Rosenmuller is on the lateral wall of the nasopharynx, just behind the cartilage of the eustachian tube.

It grows during childhood, appearing largest in size in children between 3 and 7 years of age, and begins to regress in adolescence. Children younger than 7 years are more prone to symptomatic effects of enlarged adenoid due to the relatively smaller volume of the nasopharynx and choanal opening. The prevalence of AH (pathologic enlargement) follows physiologic growth and regression pattern of the adenoid. An enlarged adenoid may block breathing and be a cause of snoring or obstructive sleep apnea. Adenoid hypertrophy can also lead to comorbid conditions such as serous otitis and sinusitis. AH is higher in frequency in children with allergic diseases, with the most common allergen being house dust. Other risk factors noted for developing AH include cigarette smoke exposure and allergic rhinitis. In a child with these risk factors, AH should be a consideration during a routine examination. Assessing adenoidal size can be achieved initially by lateral neck radiography (LNR) and assessing adenoid-nasopharyngeal ratio (A/N ratio) which is one of the most important and most widely used criteria. Although these methods are inexpensive and available, they have limited role in the exact assessment of areas such as the ears. Flexible nasal endoscopy, where adenoid size grading is on a scale of I to IV identifies the percentage of the posterior choana blocked by the adenoid tissue, with grade IV representing the highest level of obstruction.

AH influence on the pathogenesis of OME is two-fold: it may mechanically obstruct the Eustachian tube, and its vegetation may serve as a reservoir of biofilm forming bacteria causing retrograde infections towards the Eustachian tube and the middle ear.

Otitis media with effusion (OME) is a disease defined by persistence of serous or mucous fluid in middle ear without signs of an acute infection. It is amongst the most common pediatric diseases and the most common cause of hearing loss in children. It is estimated that more than 50% of children are diagnosed with OME by the age of 1 year, and up to 90% of children by the time they have reached school age.

Although the exact pathogenesis of OME is not clearly understood, it is generally resulted from lymphoid tissue overgrowth in nasopharynx, chronic sinus infection, and allergies.

It is accepted that adenoid hypertrophy (AH) is related to OME incidence. Better understanding of the correlation between the relative size of AH and the incidence of persistent OME may provide evidence to support a more standardized approach to the diagnosis and treatment of OME.

It is accepted that adenoid hypertrophy (AH) is related to OME incidence. Better understanding of the correlation between the relative size of AH and the incidence of persistent OME may provide evidence to support a more standardized approach to the diagnosis and treatment of OME.

There is sufficient evidence that AH is an important co-factor in the development of OME, a very consequential disease.

ELIGIBILITY:
Inclusion Criteria:

* Children (until age of 16 years old).
* Patients with adenoid hypertrophy.
* Patients with OME.

Exclusion Criteria:

* Children known to have cleft palate, submucous cleft palate or other medical problems causing velopharyngeal insufficiency.
* Down's syndrome, septal deviation, primary ciliary dyskinesia (Kartagener's syndrome), previous head or ear trauma, or previous myringotomy with ventilation tube insertion
* Systemic medical problems interfering with surgery.
* Refusal of parents to participate.
* Craniofacial abnormalities.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children age group (from 1 year old till 16 years old), male and female are included, with symptoms and signs of adenoid hypertrophy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Comparing presence of middle ear effusion in relation to site and size of adenoid hypertrophy | Baseline
  The incidence of OME with each AH grade occurring in each age group of the sample size.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Ahmed Salem, Professor, Study Director — Assuit University hospital

REFERENCES:
- [Background] Mnatsakanian A, Heil JR, Sharma S. Anatomy, Head and Neck: Adenoids. 2023 Jul 24. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK538137/ PMID 30844164
- [Background] Khadgi A, Koirala K, Maharjan S, Chalise K, Dhungana I, Babu Karki B. Correlation of Conductive Hearing Impairment With Sizes of Adenoids in the Pediatric Age Group: An Observational Case-Control Study. Cureus. 2023 Aug 31;15(8):e44439. doi: 10.7759/cureus.44439. eCollection 2023 Aug. PMID 37791228
- [Background] Niedzielski A, Chmielik LP, Mielnik-Niedzielska G, Kasprzyk A, Boguslawska J. Adenoid hypertrophy in children: a narrative review of pathogenesis and clinical relevance. BMJ Paediatr Open. 2023 Apr;7(1):e001710. doi: 10.1136/bmjpo-2022-001710. PMID 37045541
- [Background] Ohuche IO, Iloanusi NI, Dike CM, Chime EN. Clinical presentation, radiographic findings, and treatment outcomes in children with adenoid hypertrophy in a paediatric outpatient clinic in Enugu, Nigeria. Ghana Med J. 2023 Sep;57(3):204-209. doi: 10.4314/gmj.v57i3.7. PMID 38957679
- [Background] Galic MZ, Klancnik M. ADENOID SIZE IN CHILDREN WITH OTITIS MEDIA WITH EFFUSION. Acta Clin Croat. 2022 Feb;60(3):532-539. doi: 10.20471/acc.2021.60.03.25. PMID 35282481